CLINICAL TRIAL: NCT07204795
Title: Evaluation of the Effect of Preoperatively Administered Oral Clear Carbohydrate-Rich Drink on ObsQoR-10 Recovery Scores of Patients Undergoing Elective Cesarean Section With Neuraxial Anesthesia: A Prospective, Randomized, Controlled, Double-Blind Study
Brief Title: Effect of Preoperative Oral Carbohydrate Drink on ObsQoR-10 Score After Elective Cesarean Under Neuraxial Anesthesia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Aysenur Dostbil, Professor Dr., Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: B.30.2.ATA.0.01.00/331
Record Dates: First submitted 2025-05-17; First posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: ObsQor-10; Cesarean Section; Preoperative Fasting
Keywords: ObsQor-10; Cesarean Section; Neuraxial Anesthesia; Preoperative Fasting; Oral Clear Carbohydrate Drink

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Sham Comparator): Control Group will receive distilled water.
  Interventions: Other: Distilled water group
- Intervention Group (Experimental): This arm of patients will receive clear carbohydrate drink.
  Interventions: Other: Carbohydrate Drink

INTERVENTIONS:
Other: Distilled water group — Group A participants will receive 400 mL of distilled water orally, two hours before surgery.
  Arms: Control Group
Other: Carbohydrate Drink — Group A participants will receive 400 mL of a commercially available clear carbohydrate-rich drink orally, two hours before surgery.
  Arms: Intervention Group

SUMMARY:
The goal of this clinical trial is to determine whether a preoperative oral carbohydrate-rich clear drink can improve recovery in women undergoing elective cesarean section under neuraxial anesthesia. The main outcomes it aims to answer are:

Primary Outcome: Does the carbohydrate drink improve ObsQoR-10 scores at 24 and 48 hours postoperatively?

Secondary Outcomes: Does it reduce patients' hunger, thirst, and anxiety levels?

Researchers will compare patients receiving a 400 ml oral carbohydrate-rich clear drink 2 hours before surgery (Group A) to those receiving 400 ml distilled water (Group B), to assess differences in recovery and comfort.

Participants will:

Be randomized into two equal groups (n=50 each) using a computer-generated randomization table

Receive standardized anesthesia and postoperative analgesia

DETAILED DESCRIPTION:
This prospective, randomized, controlled, double-blind clinical trial will be conducted at Atatürk University Faculty of Medicine Hospital, following approval from the institutional ethics committee and after obtaining written informed consent from all participants. The study population will consist of 100 pregnant women scheduled for elective cesarean section under neuraxial anesthesia.Randomization will be performed using a computer-generated random numbers table by an independent statistician, allocating patients equally into two groups (Group A and Group B). Randomization will be performed using a computer-generated random numbers table by an independent statistician, allocating patients equally into two groups (Group A and Group B).

Upon arrival in the operating room, patients will undergo routine monitoring. Cesarean delivery will be performed using either spinal anesthesia or combined spinal-epidural anesthesia based on clinical indications. Intrathecal anesthesia will consist of 11.2 mg hyperbaric bupivacaine, 15 µg fentanyl, and 150 µg morphine. If additional analgesia is required through the epidural route, a mixture of 15 mL 2% lidocaine, 2 mL fentanyl, 2 mL sodium bicarbonate, and 1:200,000 adrenaline will be administered.

For intraoperative analgesia, all patients will receive 1 g intravenous acetaminophen, and, if not contraindicated, 800 mg intravenous ibuprofen. Postoperative pain management will include scheduled doses of 1 g acetaminophen and 800 mg ibuprofen every 8 hours for 48 hours. If the visual analog pain score (VAS) exceeds 3, 5 mg of oral oxycodone will be given as rescue analgesia. At discharge, patients will be prescribed up to 20 tablets of 5 mg oxycodone for breakthrough pain, with advice to continue regular acetaminophen and ibuprofen.

ELIGIBILITY:
Inclusion Criteria:

Age ≥18 years

Scheduled for elective cesarean section under neuraxial anesthesia

Gestational age ≥37 weeks

Exclusion Criteria:

Contraindication to neuraxial anesthesia

Age <18 years

Refusal to participate in the study

Obesity

Hiatal hernia

Intestinal obstruction

Gastroesophageal reflux disease (GERD)

Diabetes mellitus

Fetal anomalies

Eclampsia or preeclampsia

Substance abuse

Chronic pain conditions

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-05-20 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
ObsQor-10 Scores | From enrollment to 48th hour postoperatively
  Primary outcome assessment will be based on the ObsQoR-10 (Obstetric Quality of Recovery-10) scores at 24 and 48 hours postoperatively.

CONTACTS AND LOCATIONS:
Locations (1):
- Ataturk University Research Hospital, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Kozanhan B, Yildiz M, Polat A, Gunenc O, Tutar SM, Iyisoy MS, Kulhan NG, Sultan P. Development and Validation of a Turkish Version of Obstetric Quality of Recovery-10. Turk J Anaesthesiol Reanim. 2022 Oct;50(5):366-372. doi: 10.5152/TJAR.2022.21441. PMID 36301286
- [Background] Cho EA, Huh J, Lee SH, Ryu KH, Shim JG, Cha YB, Kim MS, Song T. Gastric Ultrasound Assessing Gastric Emptying of Preoperative Carbohydrate Drinks: A Randomized Controlled Noninferiority Study. Anesth Analg. 2021 Sep 1;133(3):690-697. doi: 10.1213/ANE.0000000000005411. PMID 33591115
- [Background] Ciechanowicz S, Setty T, Robson E, Sathasivam C, Chazapis M, Dick J, Carvalho B, Sultan P. Development and evaluation of an obstetric quality-of-recovery score (ObsQoR-11) after elective Caesarean delivery. Br J Anaesth. 2019 Jan;122(1):69-78. doi: 10.1016/j.bja.2018.06.011. Epub 2018 Jul 31. PMID 30579408